CLINICAL TRIAL: NCT05520814
Title: PD-1 Inhibitors Plus Chemoradiotherapy for Metastatic Nasopharyngeal Carcinoma: an Open-label Single-arm, Phase II Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Mei Feng, Chief Physician, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-NC-202207
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Nasopharyngeal Carcinoma; PD-1 Inhibitors; Chemoradiotherapy
Keywords: PD-1 inhibitors; concurrent; metastatic; nasopharyngeal carcinoma; chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — Immune Checkpoint Inhibitors; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- metastatic nasopharyngeal carcinoma (Experimental)
  Interventions: Drug: PD-1 inhibitors; Radiation: chemoradiotherapy

INTERVENTIONS:
Drug: PD-1 inhibitors — treprizumab injection 240mg / carrilizumab injection 200mg / Tirelizumab injection 200mg * q21d (until the disease progresses, intolerable toxicity or the investigator / subject decides to withdraw from the study, and the duration of PD-1 inhibitor is not more than 96 weeks)
Radiation: chemoradiotherapy — Chemotherapy：
  1. GP: gemcitabine 1g/m2 D1, 8 Cisplatin 80 mg/m2 d1
     * Treatment courses every 3 weeks
  2. Cisplatin 80mg/m2 d1 or carboplatin area under the curve 5mg/ml/min * Treatment courses every 3 weeks
  Radiotherapy： All the metastatic lesions received radiation dose from 30 to 60Gy according to different metastatic sites.

SUMMARY:
programmed cell death-1 (PD-1) inhibitors has been recommended as the first-line treatment for recurrent/metastatic nasopharyngeal carcinoma (R/M NPC), but progression-free survival (PFS) and overall survival (OS) was still unsatisfactory. Basic studies have already confirmed PD-1 inhibitors had concurrent synergistic effect with chemotherapy and radiotherapy. Few studies concerned about the treatment pattern for concurrent PD-1 inhibitors combination with chemoradiation for R/M NPC. There was still much uncertainties about the timing, fraction dose and total dose for PD-1 inhibitors combination with radiation. Therefore, we aimed to explore the substantial effect and toxicity of this new pattern for R/M NPC.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is one of the most common malignant tumors of the head and neck, which is derived from the epithelial cells of the nasopharynx. According to the statistics of global cancer data in 2020, there are about 129100 newly diagnosed cases of nasopharyngeal carcinoma (NPC) in the world every year, the incidence rate is less than 5 / 100000, and about 73000 people die from NPC every year. There are obvious ethnic and regional differences in the incidence of nasopharyngeal carcinoma. From the global perspective, it is more likely to occur in the yellow race, and southern China and Southeast Asia are high incidence regions of nasopharyngeal carcinoma. According to statistics, the incidence rate of nasopharyngeal carcinoma in southern China is as high as 30.29/100000 males and 13.09/100000 females. The incidence rate of male was higher than that of female. Because nasopharyngeal carcinoma is sensitive to radiotherapy and chemotherapy, and because it is adjacent to the spinal cord, brainstem, temporal lobe, optic nerve, cochlea, mandible and other important tissue structures, it cannot be treated surgically. Therefore, radiotherapy (RT) or radiotherapy combined with chemotherapy (chemotherapy) is the standard treatment for nasopharyngeal carcinoma.

Although the diagnosis and treatment of nasopharyngeal carcinoma have been greatly improved under the background of the development of imaging technology and the era of precision radiotherapy, the situation it faces is still not optimistic. On the one hand, 4% - 10% of newly diagnosed nasopharyngeal carcinoma has distant metastasis; on the other hand, about 10% of nasopharyngeal carcinoma has local and regional recurrence after intensity modulated radiation therapy (IMRT) ± chemotherapy, and 15% - 30% of patients have distant metastasis after radical treatment. Therefore, recurrence and metastasis are still the main causes of treatment failure of nasopharyngeal carcinoma. This poses a severe challenge to the treatment mode of nasopharyngeal carcinoma (NPC).

In the era of traditional treatment, surgery is the first choice for the treatment of recurrent nasopharyngeal carcinoma. The standard treatment for patients with recurrent or metastatic nasopharyngeal carcinoma (R / M NPC) that cannot be cured by surgery is platinum based dual drug palliative systemic chemotherapy. At present, the GP regimen of gemcitabine combined with cisplatin is the standard first-line treatment for R / M NPC, but the progression free survival (PFS) of first-line chemotherapy is still less than 7 months, and the median overall survival (OS) is difficult to exceed 30 months [17]. In view of the limited progress of chemotherapy drugs, we urgently need new treatment schemes to prolong the survival time of R / M NPC patients. Immunotherapy is a hot topic in R / M NPC Research in recent years, and it is expected to prolong the long-term survival of patients. Immunotherapy also has a large number of clinical studies in R / M NPC patients, making the treatment of nasopharyngeal carcinoma enter an era of immunotherapy.

The occurrence of nasopharyngeal carcinoma is related to the chronic infection of Epstein Barr virus (EBV). Nasopharyngeal carcinoma cells infected with EBV express target proteins of CD4 and CD8 positive T cells (CD4 + T and CD8 + T), and nasopharyngeal carcinoma cells infected with EBV undergo four different latent cycles (phase 0-IV). The researchers found that NPC cells expressed specific latent proteins (EBNA1, LMP1, LMP2 and lmp2b) in latent phase II. Through basic research, it was found that these four latent proteins are EBV antigens expressed by nasopharyngeal carcinoma cells, contain more CD4 + T and CD8 + T cell epitopes, and are almost only expressed in nasopharyngeal carcinoma cells. Therefore, these four latent proteins are ideal targets for immune precision therapy. On the other hand, there are a large number of tumor infiltrating lymphocytes (TILs) in tumor tissues, including a large number of CD4 + T and CD8 + T lymphocytes, which can accurately attack EBV antigens expressed by nasopharyngeal carcinoma cells. However, in patients with nasopharyngeal carcinoma with high lymphocyte infiltration, tumor cells can still continue to grow. This phenomenon indicates that there is an immunosuppressive microenvironment in nasopharyngeal carcinoma. Immunotherapy can effectively improve the immunosuppressive microenvironment, making immunotherapy more widely used in the occurrence, development and clinical diagnosis and treatment of nasopharyngeal carcinoma. Inhibitory receptors expressed by T cells, antigen-presenting cells and other cells exert corresponding immune effects after binding with their corresponding ligands, which are collectively referred to as "immune checkpoints". Among them, programmed death receptor-1 (PD-1) and its ligand programmed death ligand-1 (PD-L1) are important targets of immunotherapy.

PD-L1 (also known as CD274 and B7-H1) is a type I transmembrane protein containing 290 amino acids in the immunoglobulin superfamily, which is similar to the immunoglobulin light chain. In 1999, it was found that it is expressed in the heart, placenta, lung and skeletal muscle and regulates T cell proliferation. Through anti-T cell receptor and CD28 costimulatory signal, it binds to its main receptor PD-1 in trans and CIS, thereby inhibiting the function of anti-tumor PD-1 positive T cells. PD-L1 also interacts in cis and trans with another known receptor, the immune co signaling molecule CD80, to prevent co stimulation of T cells. PD-1 / PD-L1 pathway maintains the normal immune state of the body. In the tumor microenvironment, PD-L1 expressed or overexpressed on the surface of tumor cells binds to the PD-1 target expressed on the surface of T cells, inhibits the normal function of T cells, weakens the recognition and response ability of T cells to tumor cells, thereby realizing tumor immune escape and forming an immunosuppressive microenvironment. In short, the main anti-tumor mechanism of PD-1 / PD-L1 inhibitors is to block PD-1 and its ligand PD-L1, which are involved in attenuating the activation pathway of T cells, and prevent or reverse the acquired peripheral tolerance to tumor antigens, thus leading to T cell recovery, reducing T cell failure or death, increasing T cell memory and anti-tumor immune cell infiltration in tumors, enhancing T cell activity, playing an anti-cancer role, and significantly prolonging the survival of patients. Some researchers further found that PD-L1 overexpression was common in NPC patients, which may be related to EBV infection. Comprehensive analysis shows that there are a large number of immune cells in NPC tissues, but due to EBV infection and other reasons, NPC cells overexpress PD-L1, resulting in immunosuppressive effect. The use of PD-1 immune checkpoint inhibitors can theoretically reactivate the immune response, so that lymphocytes infiltrating the tumor microenvironment of nasopharyngeal carcinoma can play an immune role, and ultimately achieve the goal of tumor suppression. Immunotherapy based on PD-1 / PD-L1 immune checkpoint inhibitors has made a breakthrough in the treatment of nasopharyngeal carcinoma. At present, many studies on anti-PD-1 monoclonal antibody in nasopharyngeal carcinoma have been officially published.

Keynote-028 study is a non randomized, multicenter phase I and B clinical trial to explore the efficacy and safety of pembrolizumab in patients with PD-L1 positive nasopharyngeal carcinoma. Twenty seven NPC patients with PD-L1 expression who could not be operated or distant metastasis and failed standard treatment were included in the study. The median follow-up time was 20 months, the objective response rate (ORR) was 25.9%, the median PFS was 6.5 months, and the median OS was 16.5 months. PD-L1 expression had a certain correlation with the treatment effect. The incidence of drug-related adverse events (AES) was 74.1%, and the incidence of grade 3-5 AES was 29.6%. This study showed that pabilizumab showed strong antitumor activity and manageable safety in pd-l1-positive recurrent / metastatic nasopharyngeal carcinoma. Similar to pabolizumab, the nci-9742 study is a single arm, multicenter phase II clinical study on nivolumab. 44 patients with nasopharyngeal carcinoma who progressed after the treatment of advanced platinum containing regimen were enrolled in the study, and received the single drug treatment regimen of nabulizumab. The final results showed that 1 patient obtained Cr, 8 patients obtained pr (ORR 20.5%), the 1-year OS rate was 59%, and the tolerance was good. The results of the study confirmed that the monotherapy of nabulizumab may be effective and safe for advanced nasopharyngeal carcinoma.

At present, PD-1 monoclonal antibody has shown a certain efficacy in patients with recurrent / metastatic nasopharyngeal carcinoma. The median PFS of immunomonotherapy used in the posterior line treatment of R / M NPC is mostly 3-4 months, and the median OS is concentrated in 16-17 months. The overall incidence of side effects is lower than that of chemotherapy, and it is well tolerated. It can bring longer survival benefits for patients, but the benefit population is small (20% - 30%).

In 2021, the cancer prevention and treatment center of Sun Yat sen University led two phase III, double-blind, randomized controlled clinical studies of immunotherapy combined with gemcitabine and cisplatin (GP) chemotherapy for advanced first-line nasopharyngeal carcinoma: captain-1st study and jupiter-02 study. Captain-1st study [45] confirmed that in the first-line treatment of locally recurrent or metastatic nasopharyngeal carcinoma, carrilizumab combined with GP chemotherapy was used for the first-line treatment of R / M NPC, with a median PFS of 10.8 months, an orr of 88.1%, a median duration of remission (DOR) of 9.9 months, and good safety. The jupiter-02 study [46] confirmed that in the first-line treatment of locally recurrent or metastatic nasopharyngeal carcinoma, the first-line treatment of R / M NPC with treprizumab combined with GP chemotherapy had a median PFS of 11.7 months, HR of 0.52, and median dor of 10.0 months. The risk of death was reduced by 40%, and the safety was good. These two studies confirmed that although the adverse reactions of chemotherapy combined with PD-1 mAb were different compared with the placebo group, the overall safety was controllable.

Compared with PD-1 inhibitor immunomonotherapy, PD-1 monoclonal antibody combined chemotherapy can bring longer survival benefits to patients in the treatment of recurrent / metastatic nasopharyngeal carcinoma, obtain better treatment effect and controllable safety. However, some patients still have poor treatment effect, with an effective rate of about 50%, which poses a severe challenge to the era of immunotherapy for recurrent / metastatic nasopharyngeal carcinoma.

At present, a large number of basic studies have confirmed that PD-1 inhibitors have synergistic effects with radiotherapy. Radiotherapy can stimulate the immune response, promote the death of immunogenic cells and release tumor associated antigen (TAA), and enhance the homing of immune cells to tumors, thus transforming immunologically "cold" tumors into "hot" tumors. In addition, radiotherapy induces an increase in PD-L1 expression on tumor cells, making them more susceptible to continuous effects of PD-1 / PD-L1 inhibitors, thus promoting longer survival time and higher response rate. In addition, radiotherapy may cause distant effect, shrink the target tumor outside the radiation field area, and may also increase the aggregation of T cells in the tumor microenvironment, promote cytokine secretion and antigen presentation.

Recently, Professor Chen Mingyuan from the cancer prevention and treatment center of Sun Yat sen University led an open, single arm, phase II clinical study to explore the efficacy and safety of treprizumab combined with intensity modulated conformal radiotherapy (IMRT) in the treatment of recurrent nasopharyngeal carcinoma (rnpc) [63]. In this study, 25 patients with unresectable rnpc were included. All patients received treprizumab combined with IMRT, with a median IMRT dose of 60.21 Gy. The results showed that after 3 months of radiotherapy, the objective response rate (ORR) was 79.2% and the disease control rate was 95.8% in 24 evaluable patients. The median PFS was 18.67 months, the 12-month PFS rate was 91.8%, and the median OS was not reached. In terms of safety, the most common adverse events (AES) were all grade 1-2, and the safety was manageable. It has been proved that treprizumab combined with IMRT showed promising antitumor activity in patients with recurrent nasopharyngeal carcinoma, achieved good remission rate and PFS outcome, and was well tolerated.

At present, PD-1 inhibitor immunomonotherapy or combined chemotherapy has been widely used in patients with recurrent / metastatic nasopharyngeal carcinoma, and it is also the first-line treatment for R / M NPC recommended by international and domestic guidelines. However, few studies have focused on the simultaneous combination of PD-1 inhibitors and chemoradiotherapy. More trials are needed to explore the possibility of combining PD-1 inhibitors with chemoradiotherapy, which may be a new treatment strategy for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the trial and sign the informed consent for the study in writing.
2. Age ≥ 18 years old (when signing the informed consent for this study).
3. Metastatic disease after primary standard treatment (patients who had metastatic diseases over six months after treatment)
4. Metastatic lesions are not suitable for surgery.
5. According to recist1.1 evaluation criteria, there are measurable lesions (1-5 measurable lesion).
6. The physical state of the Eastern Cooperative Oncology Group (ECoG) was 0-1.
7. Tumor tissue can be provided for PD-L1 expression detection: newly obtained biopsy (within 90 days before the start of study treatment) is preferred. If biopsy tissue cannot be provided for detection, archived tissue wax block can be provided for post-section detection.
8. Urine pregnancy test was negative (female), and contraceptive measures were taken from the trial period to 3 months after the end of the trial.
9. The function of main organs is normal, and the blood routine examination shall meet the following standards: WBC ≥ 4.0 × 109/L，ANC≥2.0 × 109/L， PLT≥100 × 109 / L, Hb ≥ 90g / L (no blood transfusion and blood products within 14 days, no correction with G-CSF and other hematopoietic stimulating factors); Biochemical examination shall meet the following standards: TBIL ≤ 2.0 × ULN，ALT、AST≤2.5 × ULN, bun and cre ≤ 1.5 × The clearance rate of ULN or endogenous creatinine ≥ 60ml / min (Cockcroft Gault formula); Good coagulation function: defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; If the subject is receiving anticoagulant treatment, as long as Pt is within the proposed scope of use of anticoagulant drugs; The myocardial enzyme spectrum was within the normal range.
10. According to the judgment of the investigator, the patient was considered to be able to comply with the protocol.

Exclusion Criteria:

1. Locally advanced nasopharyngeal carcinoma has disease progression (PD) within 6 months after systemic treatment.
2. It is known that any component of the investigational drug or preparation has caused severe hypersensitivity, including severe hypersensitivity to other monoclonal antibodies, gemcitabine, taxol, fluorouracil, platinum and other related compounds (NCI ctcaev5.0 ≥ grade 3).
3. According to the criteria of common adverse event terminology (NCI ctcaev5.0), there were peripheral neuropathy ≥ grade 2.
4. Other malignant tumors occurred within 5 years or present at the same time.
5. Interstitial lung disease or non communicable pneumonia (including past history and present condition); Local interstitial pneumonia induced by radiotherapy is excluded.
6. Have uncontrolled systemic diseases, including diabetes, hypertension, acute lung disease, etc.
7. Active infections requiring systemic treatment, including active tuberculosis.
8. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage.
9. There are obvious cardiovascular diseases, heart failure classified as grade 2 or above by the New York Heart Association (NYHA), previous myocardial infarction within 3 months, unstable arrhythmia (including QT interval ≥ 480 MS) or unstable angina pectoris.
10. Active central nervous system metastasis and / or cancerous meningitis (before the first administration, except for patients with stable brain metastases: subjects with brain metastases who have received previous treatment can participate in the study, provided that they are clinically stable for at least 2 weeks, there is no evidence of new or expanded brain metastases, and steroids are stopped 3 days before the administration of the study drug. Except for subjects with asymptomatic brain metastases: they have no neurological symptoms, do not need corticosteroids, and have no lesions > 1.5cm, and they need regular brain tests as disease sites Imaging examination.)
11. Active hepatitis B or C, meeting any of the following conditions: hepatitis B virus deoxyribonucleic acid (HBV DNA) in peripheral blood is positive (the result is greater than the detection limit of the analysis method); Hepatitis C virus RNA (HCV RNA) in peripheral blood was positive (the result was greater than the detection limit of the analysis method).
12. Patients with a history of immune deficiency, including HIV positive and / or other acquired and congenital immune deficiency diseases, and / or patients with a history of organ transplantation.
13. Active autoimmune diseases that may worsen when receiving systemic steroid therapy or any other form of immunosuppressive therapy (except for patients with type I diabetes, vitiligo, psoriasis or hypothyroidism or hyperthyroidism that do not require immunosuppressive therapy).
14. Immunosuppressive drugs are used, except for the following cases: intranasal, inhaled, topical steroids or local steroid injections (e.g., intra-articular injections), physiological doses of systemic corticosteroids (≤ 10 mg / day prednisone or equivalent dose), steroid pre medication for hypersensitivity reactions (e.g., CT scan pre medication).
15. Major surgery was performed within 4 weeks before enrollment, and / or there were unhealed wounds, ulcers or fractures.
16. Live virus vaccine (seasonal influenza vaccine and coronavirus vaccine without live virus are allowed to be inoculated) was inoculated within 4 weeks before enrollment.
17. Currently participate in and receive research treatment, or participate in research drug trials and receive research treatment or use research devices within 4 weeks before enrollment.
18. Patients with known drug abuse and / or psychosis have severe intellectual or cognitive impairment, which may interfere with the cooperation with the trial requirements.
19. Pregnancy, lactation, and / or expected pregnancy or childbirth during the trial period, from the beginning of the screening visit to 180 days after the last dose of study drug.
20. Anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibodies and / or any other antibody or drug specifically targeting T cell costimulation or immune checkpoint pathway.
21. patients who cannot follow the trial protocol or cooperate with follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3 months post radiotherapy
  Three months after the end of radiotherapy, the proportion of patients whose tumors shrink to a certain amount and remain for a certain time, including those with complete remission (CR) + partial remission (PR).

SECONDARY OUTCOMES:
overall survival (OS) rate | 1, 2-year
  1, 2-year overall survival (OS) rate
Progression-free survival (PFS) rate | 1,2-year
  1, 2-year Progression-free survival (PFS) rate
Disease Control Rate(DCR) | 3 months post radiotherapy
  Three months after the end of radiotherapy, the proportion of patients whose tumors shrink to a certain amount and remain for a certain time, including those with complete remission (CR) + partial remission (PR)+Stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China